CLINICAL TRIAL: NCT04587141
Title: Impatto Clinico Dell'Anemia Nelle Malattie Infiammatorie Intestinali: Ruolo Della Carenza di Ferro e Della Terapia Sostitutiva Con Ferro, Trial Terapeutico (RIDART II)
Brief Title: Clinical Burden of Anemia in Inflammatory Bowel Disease: Therapeutic Trial
Acronym: RIDARTII
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Collaborators: Italian Group for the study of Inflammatory Bowel Disease (IG-IBD) (Other)
Responsible Party: Principal Investigator, Antonio Di Sabatino, Professor, Fondazione IRCCS Policlinico San Matteo di Pavia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRCCSPSM 2
Record Dates: First submitted 2020-10-07; First posted 2020-10-14 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Iron Deficiency Anemia; Inflammatory Bowel Diseases
Keywords: anemia; iron deficiency; Crohn's disease; Ulcerative colitis
MeSH Terms: conditions — Anemia, Iron-Deficiency; Inflammatory Bowel Diseases; Anemia; Iron Deficiencies; Crohn Disease; Colitis, Ulcerative | interventions — sucrosomial iron; ferric gluconate; ferric carboxymaltose

STUDY DESIGN:
Intervention Model Description: Three iron supplementation regimens will be compared in terms of effectiveness and safety in the treatment of IBD-associated IDA. Primary outcome is the relative effectiveness of an oral iron supplementation regimen compared with two iv iron regimens.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Sucrosomial iron (Experimental): One or two capsules/die of sucrosomial iron will be assumed by the participant, depending on hemoglobin (Hb) concentration and participant body weight, for 8 weeks. Each capsule contains 30 mg of iron.
  Interventions: Drug: Sucrosomial iron
- Ferric gluconate (Active Comparator): Ferric gluconate will be administered by iv infusion, 125 mg of elemental iron once or twice weekly for 4 or 8 weeks depending on Hb concentration and patient body weight.
  Interventions: Drug: Ferric Gluconate
- Ferric carboxymaltose (Active Comparator): Two or three iv infusions of 500-1000 mg of elemental iron will be given as ferric carboxymaltose, over a 4 week period. Dosage and number of infusions will be established depending on Hb concentration and patient body weight.
  Interventions: Drug: Ferric carboxymaltose

INTERVENTIONS:
Drug: Sucrosomial iron — This is an oral iron formulation commercially available as an integrator
  Other Names: Sideral
  Arms: Sucrosomial iron
Drug: Ferric Gluconate — This is a commercially available iron formulation for parenteral administration
  Other Names: Ferrlecit
  Arms: Ferric gluconate
Drug: Ferric carboxymaltose — This is a commercially available iron formulation for parenteral administration
  Other Names: Ferinject
  Arms: Ferric carboxymaltose

SUMMARY:
Anemia is the most common extraintestinal manifestation of inflammatory bowel diseases (IBD), Although most cases of anemia in IBD are due to iron deficiency, many patients with iron deficiency anemia (IDA) are not treated with iron supplementation. In addition, it has not been firmly established which iron supplementation modality provides the best results in terms of effectiveness and safety. In the present study the investigators will compare the effectiveness and efficacy of three iron supplementation modalities in IBD-associated IDA. There will be two arms of parenteral (iv) iron supplementation (ferric carboxymaltose and ferric gluconate) and one arm of oral supplementation (sucrosomial iron). Primary objective of the study is is to compare the efficacy of oral iron with that of the iv iron supplementation regimens. The primary outcome is measured as the percentage of patients responsive to iron supplementation. Response is defined by Hb normalization or by an Hb increase ≥2 g/dL by week 8 from start of therapy. As secondary objectives the influence of anemia and its treatment on fatigue, quality of life, hospitalizations, additional outpatient visits, number of endoscopic examinations; further treatments and relative side effects will be evaluated.

DETAILED DESCRIPTION:
Anemia is the most common extraintestinal manifestation of inflammatory bowel diseases (IBD). Most cases of anemia in IBD are due to iron deficiency (IDA) and to anemia of inflammation (AI) (Bergamaschi et al, 2010). Guidelines by the European Crohn's and Colitis Organisation (ECCO) suggest that iron supplementation should be started when IDA is present or even in the presence of iron deficiency without anemia (Dignass et al, 2015). However, many IBD patients with IDA are not properly treate, probably due to the belief that mild to moderate degrees of anemia may not have a significant impact on the patient's quality of life, that oral iron supplementation may adversely affect disease activity, and that parenteral iron administration may cause severe side effects. In this study the investigators will compare three iron supplementation regimens (two iv iron formulations and one oral iron integrator) for the treatment of IDA in patients with IBD in terms of both efficacy and safety. Participation to the trial does not involve additional risks for the patients. In fact, the trial does not require additional diagnostic procedures beyond those that are usually performed in IBD patients and the drugs that will be use din the trial are already used in patients with IBD and IDA. According to WHO criteria (WHO scientific groupl, 1968), anemia is defined as Hb <13.0 g/dL in males and Hb <12 g/dL in females (Blanc et al, 1968). A serum ferritin <30 µg/L or a serum ferritin ≤100 µg/L with transferrin saturation <20% are required for the diagnosis of isolated IDA and of IDA associated with inflammation, respectively.

300 subjects with IDA and IBD will be recruited in a multicenter trial and randomized 1:1:1 to the three iron replacement arms. Expected duration of subject participation to the trial will be 24 weeks for each patient, consisting of an 8 week treatment period, with follow-up visits at weeks 4, 8, 12 and 24 from treatment start.

Study participants can be participating in other research, either observational or interventional, or other drug research concerning the treatment of IBD.

Iron gluconate and FCM are licensed for use in Italy and will be used according to AIC. Iron gluconate will be part of the normal hospital stock. FCM will be purchased through an IG-IBD donation to the Fondazione IRCCS Policlinico San Matteo. Microsomial iron is a formulation for oral administration commercially available in Italy as an iron integrator; for the study, however, it will be provided free of charge from Pharmanutra S.r.l.

Concomitant therapy No other iron supplementation is allowed during the trial. Vitamin integrators containing folic acid, vitamin B12 and vitamin D or calcium are allowed, as well as any other treatment for IBD and related comorbidities; therefore, study patients can be treated with topic and systemic mesalazine and steroids, or with immunosuppressors (azathioprine, mercaptopurine, cyclosporine, methotrexate) and biologic immunomodulators (infliximab, adalimumab, golimumab) commonly used in IBD patients; pain relievers and antibiotics (the latter for either infection treatment or profilaxis) can be used without restrictions.

Procedures and assessments Laboratory assessments can be performed outside the participating Centers, and results faxed or emailed to the Investigators who will register data in the eCRF. Result notification to the trial team must be performed as soon as possible.

Safety/Adverse events (AE)/Serious AE (SAE) review as well as treatment compliance review at scheduled time points will be included during every visit. This will be included specifically in the list of assessments.

Subject Registration Subjects will be registered locally and assigned a registration number/code. This number, together with the Center code, will constitute the unique patient identification code. Only the patient physicians must be able to identify the patient from the assigned code. Randomization will be performed by the Coordinator Center.

Baseline assessments

All patients will have a full medical history taken and a clinical examination. The following data points are to be recorded:

a) Weight in Kg b) Gender c) Age (year of birth) d) Any significant past medical history e) CDAI and CAI disease activity scores for CD and UC respectively f) Full blood count (including platelets and differential white cell count) g) Biochemical series: including creatinine, serum iron, transferrin, serum ferritin, C reactive protein (PCR), folic acid, vitamin B12 and urine pregnancy test for women of childbearing potential (these are mandatory tests; further biochemical parameters useful for the study are reported in the CRF) h) Tests for HIV, HCV, HBsAg, QuantiFERON TB-2G (QuantiFERON is not necessary in patients previously treated for latent or active TB as per local standard of care) i) IBDQ score, VAS evaluation of fatigue J) Actual treatment k) Chest radiograph l) A blood sample (two 1.5 mL serum vials) will be obtained and stored at -20° C.

Timing of assessments Follow-up will be performed at weeks 4, 8, 12 and 24.

The following data are to be recorded:

1. Physical examination
2. Adverse Event Review
3. Weight in Kg

e) Full blood count f) Biochemical series g) IBDQ score, VAS evaluation of fatigue h) Actual treatment i) One blood sample (two 1.5 mL serum vials) will be obtained at the week 8 follow-up visits and stored at -20° C.

Long-Term Follow-up Assessments After the end of the study patients will be followed-up as usual for their conditions. Telephone calls will be used to contact patients if visits or data collection time-points are missed; whenever data collection will be impossible, the patient will be identified as 'lost to follow-up'.

Patients will be expected to return to normal standard of care following their participation in the trial.

Trial restrictions

Women of childbearing potential participating in the trial are required to use adequate contraception for the duration of the trial and for 3 months after the completion of the trial/last treatment. This includes:

* Intrauterine Device (IUD)
* Hormonal based contraception (pill, contraceptive injection or implant etc)
* Barrier contraception (condom and occlusive cap e.g. diaphragm or cervical cap with spermicide)
* True abstinence (where this is in accordance with the patients preferred and usual lifestyle)
* Men are not required to use contraception and do not need to refrain from donating sperm for the duration of the trial and any period thereafter.

Assessment of efficacy will be performed at 4, 8, 12 and 24 weeks after the start of treatment and will be based on determination of complete blood counts. Other informations concerning laboratory parameters, quality of life, clinical course, serum hepcidin and inflammatory cytokine concentrations will be gathered at the scheduled follow-up visits.

Data analysis Primary endpoint: the rate of response will be compared between groups with the Fisher exact test. The combined iv regimens will be compared to the oral regimen at the 5.0% significance level. Difference in response rate (iv regimens - oral regimen) and 95% confidence interval will be computed. If the lower limit of the confidence interval for the difference in rates is above 15%, the non-inferiority limit, non-inferiority will be claimed. If non inferiority is shown overall, 97.5% confidence intervals will be computed for the difference of oral vs each i.v. regimen and non-inferiority will be assessed as above. Finally if non inferiority against the combined iv regimen is shown, superiority will be tested at the same 5% level.

Further paired comparisons will be performed using the Bonferroni correction and will be considered descriptive only.

The primary endpoint will be analyzed both in the intention to treat and in the per-protocol (PP) population. In a non inferiority setting. The PP population represents the primary population.

Data handling and record keeping All data will be transferred into an electronic Case Report Form (eCRF) identified by a patient code. All trial data in the eCRF will be extracted from and be consistent with the relevant source documents. The eCRFs will be completed, dated and electronically signed by the investigator or designee in a timely manner. It remains the responsibility of the investigator for the timing, completeness and accuracy of the eCRF pages. The eCRF will be accessible to trial coordinators, data managers, the investigators, Clinical Trial Monitors, Auditors and Inspectors as required. The investigator will maintain a logbook with patients identification and the allocated codes in the investigator study file.

Remote data-entry will be performed through the RedCap platform by each investigator. A paper copy of the eCRF will be provided with the investigator study file.

Remote monitoring of the eCRF completeness and incongruences will be performed at the clinical trial center of the coordinating center and queries will be submitted to the investigators as appropriate.

The investigator will also supply the trial coordination Center with any required, background information from the medical records as required. Data should be entered into the database within 2 months of the patient visit being completed.

The investigators may retain copies of the eCRF in the relevant sections of their Investigator Site File with any required coded background information from the medical records as required.

Source Data The investigators agree to keep records of all participating patients: sufficient information to link eCRFs, hospital records and samples, all original signed informed consent forms and copies of the CRFs, Patient Medical Records, On-line test results, sample logs.

Data Safety Monitoring Board/Trial Steering Committee The study has been planned in Pavia by Prof. A. Di Sabatino, Dr. G. Bergamaschi and Prof. G.R. Corazza, from the Department of Internal Medicine, and DR. C. Klersy, Servizio di Biometria, all from Fondazione IRCCS Policlinico San Matteo; they represent the Trial Steering Committee.

Consent The Informed Consent is in compliance with GCP, local regulatory requirements and legal requirements. Informed consent from each patient or the patient's legally acceptable representative will be obtained before any trial-specific activity is performed. The informed consent form used and any change made during the course of this trial, will be submitted to the REC. The investigator will retain the original of each patients signed informed consent form.

Should a patient require a verbal translation of the trial documentation by a locally approved interpreter/translator, it is the responsibility of the individual investigator to use locally approved translators.

Any new information which becomes available, which might affect the patient's willingness to continue participating in the trial, will be communicated to the patient as soon as possible. This may occur either verbally over the telephone, or at their next visit (if visits are close together).

Regulatory Compliance The trial started after approval by the National Competent Authority and by the Ethics Committees of the participating Centers. The protocol and trial conduct will comply with the Medicines for Human Use (Clinical Trials) Regulations 2004.

The trial will be performed in accordance with the spirit and the letter of the declaration of Helsinki, the conditions and principles of Good Clinical Practice, the protocol and applicable local regulatory requirements and laws.

Sponsorship, Financial and Insurance The trial has obtained financial support from IG-IBD for patients' insurance, FCM procurement and FCM and microsomial iron shipment to participating Centers. Microsomial iron will be provided for free from Pharmanutra S.r.l.

ELIGIBILITY:
Inclusion Criteria:

To be included in the trial the patient must:

* Have given written informed consent to participate
* Be aged 18 years and over
* Have a BMI >16
* Have IBD and IDA with or without inflammation

Exclusion Criteria:

* Patients with hypersensitivity to the IMPs, to other iron containing products and to sucrose or benzil alcohol will be excluded from the study.

  * Pregnancy, lactation and women of childbearing potential (WOCBP) (i.e. fertile, following menarche and until becoming post-menopausal, no menses for 12 months without an alternative medical cause, unless permanently sterile) that are not willing to use highly efficient contraceptive measures according to the CTFG recommendations on contraception (Table 4);
  * male patients with WOCBP partners who are unwilling to use highly efficient contraceptive measures (Table 4);
  * an history of erythropoietin treatment within 4 weeks prior to recruitment;
  * alcohol abuse, liver cirrhosis, active hepatitis or signs of liver disease with a Child-Pugh class B or C;
  * chronic renal failure stage 3 or higher (estimated glomerular filtration rate <60mL/min as determined using either the CKD-EPI equation, the MDRD equation or the Cockcroft-Gault formula);
  * major surgery in the previous 3 months;
  * significant overt bleeding, acute severe anemia with hemodynamic instability;
  * active malignancy and any hematologic disease causing anemia;
  * known active infection;
  * known human immunodeficiency virus HCV and HBV infections;
  * evidence of tubercular (TB) infection (see section 5.2.1 for the TB screening criteria necessary to rule out active or latent TB infection).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Relative efficacy of the three iron supplementation regimens | The primary outcome will be measured at week 8 from start of iron supplementation
  Primary endpoint of the trial is to compare the efficacy of oral iron with that of the iv iron supplementation regimens in the treatment of IDA in IBD. The primary comparison of interest regards the 2 combined iv regimens vs. the oral iron supplementation. Non inferiority of the oral regimen is hypothesized. Primary outcome measure is the proportion of patients responsive to iron supplementation. Response is defined by Hb normalization or by an Hb increase ≥2 g/dL by week 8. Normalization of Hb occurs with Hb values ≥12 g/dL in females or ≥13 g/dL in males.

SECONDARY OUTCOMES:
Safety evaluation: Adverse events | Enrollment to 24 weeks
  Adverse events will be registered. Severe adverse events will be reported to the competent Authorities
Influence of anemia and its treatment on fatigue | Enrollment to 24 weeks
  Fatigue will be measured through a Visual Analogue Scale (VAS) at patient recruitment and at the scheduled follow-up visits. The range of the visual scale is from 0 to 100, with higher scores indicating more severe fatigue
Evaluation of quality of life | Enrollmen to to 24 weeks
  Quality of life will be measured using the italian validated version of the Inflammatory Bowel Disease Questionnaire (IBDQ, Ciccocioppo et al, 2011)
Number of hospitalizations, additional outpatient visits, number of endoscopic examinations, further treatments | Enrollment to 24 weeks
  number of hospitalizations, additional outpatient visits, number of endoscopic examinations, further treatments and their relation with treatment and anemia degree will be determined.

OTHER OUTCOMES:
Serum Hepcidin | 8 weeks
  Serum hepcidin concentration (ng/mL) will be determined at recruitment and at the end of the iron supplementation period.
Serul IL-6 | Enrollment
  Serum concentration of IL-6 (pg/mL) will be determined at patient recruitment
Serum IL-1 beta | Enrollment
  Serum concentration of IL-1 beta (pg/mL) will be determined at patient recruitment
Serum TNF-alpha | Enrollment
  Serum concentration of TNF-alpha (pg/mL) will be determined at patient recruitment

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Di Sabatino, MD, Principal Investigator — Fondazione IRCCS Policlinico San Matteo di Pavia
Locations (1):
- Fondazione IRCCS Policlinico San Matteo, Pavia, Italy

IPD SHARING:
Plan to Share IPD: No
Individual participant data will be available to other researchers upon request.

REFERENCES:
- [Background] Nutritional anaemias. Report of a WHO scientific group. World Health Organ Tech Rep Ser. 1968;405:5-37. No abstract available. PMID 4975372
- [Background] Dignass AU, Gasche C, Bettenworth D, Birgegard G, Danese S, Gisbert JP, Gomollon F, Iqbal T, Katsanos K, Koutroubakis I, Magro F, Savoye G, Stein J, Vavricka S; European Crohn's and Colitis Organisation [ECCO]. European consensus on the diagnosis and management of iron deficiency and anaemia in inflammatory bowel diseases. J Crohns Colitis. 2015 Mar;9(3):211-22. doi: 10.1093/ecco-jcc/jju009. Epub 2014 Dec 3. No abstract available. PMID 25518052
- [Background] Ciccocioppo R, Klersy C, Russo ML, Valli M, Boccaccio V, Imbesi V, Ardizzone S, Porro GB, Corazza GR. Validation of the Italian translation of the Inflammatory Bowel Disease Questionnaire. Dig Liver Dis. 2011 Jul;43(7):535-41. doi: 10.1016/j.dld.2010.12.014. Epub 2011 Feb 18. PMID 21315666
- [Background] Bergamaschi G, Di Sabatino A, Albertini R, Ardizzone S, Biancheri P, Bonetti E, Cassinotti A, Cazzola P, Markopoulos K, Massari A, Rosti V, Porro GB, Corazza GR. Prevalence and pathogenesis of anemia in inflammatory bowel disease. Influence of anti-tumor necrosis factor-alpha treatment. Haematologica. 2010 Feb;95(2):199-205. doi: 10.3324/haematol.2009.009985. Epub 2009 Oct 8. PMID 19815838
- See also: RIDART studies site — https://sites.google.com/site/ridartstudy/
- See also: RIDART I study site — https://sites.google.com/site/ridartstudy/home/ridart-ii